CLINICAL TRIAL: NCT05126823
Title: Efficacy of a Combined Acceptance and Commitment Intervention to Improve Psychological Flexibility and Associated Symptoms in Cancer Patients: a Randomized Controlled Clinical Trial
Brief Title: Efficacy of a Combined ACT+ App Intervention to Improve Psychological Flexibility and Associated Symptoms in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Garcia Torres (Other)
Responsible Party: Sponsor-Investigator, Francisco Garcia Torres, Lecturer, Universidad de Córdoba
Organization: Universidad de Córdoba (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PY20_00485
Record Dates: First submitted 2021-10-27; First posted 2021-11-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Cancer; Oncology; Acceptation and commitment therapy; Psychological flexibility; Randomized controlled trial
MeSH Terms: conditions — Neoplasms | interventions — Amyloid; Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: This study is a three-arm randomized clinical trial, with a pre-post-follow-up repeated measures intergroup design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ACT face-to-face + app (Experimental): Combines face-to-face ACT sessions with non-face-to-face activities and resources (mobile applications)
  Interventions: Behavioral: Acceptance and commitment therapy + app
- ACT face-to-face (Active Comparator): face-to-face ACT sessions
  Interventions: Behavioral: Acceptance and commitment therapy
- Waitlist (No Intervention): Waitlist group. After the second assessment of the two ACT groups (at post-treatment) this group will receive the face to face ACT intervention.

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy + app — In the group ACT+app, experiential exercises are carried out, metaphors, discussions and assignments are used to promote awareness and flexibility about the thoughts and emotions associated with cancer and interleaved non-contact activities, which will serve as support for each of the modules. The non-contact activities will consist of assigning tasks, practices (mindfulness, breathing), reminder systems, recording, reinforcement and monitoring. Resources such as short texts, videos, audio files and recording systems will be used
  Arms: ACT face-to-face + app
Behavioral: Acceptance and commitment therapy — In the group ACT, experiential exercises are carried out, metaphors, discussions and assignments are used to promote awareness and flexibility about the thoughts and emotions associated with cancer
  Arms: ACT face-to-face

SUMMARY:
Introduction: emotional and physical alterations frequently appear in cancer patients. In this sense, interventions based on acceptance and commitment therapy (ACT) show their efficacy to improve these symptoms through increased psychological flexibility, however, there is little evidence of the efficacy of ACT using combined modality (face-to-face + app), despite the fact that this application modality may have beneficial effects in this group of patients, who may see their participation in the interventions limited as a consequence of the disease.

Method / design: Cancer patients will be randomly assigned to one of the following groups: (1) face-to-face ACT + app group, (2) face-to-face ACT group, and (3) group receiving usual treatment. The planned interventions last between 8 and 10 weeks and include experiential exercises, metaphors, discussions, and homework assignments to promote awareness and flexibility about thoughts and emotions associated with cancer. In the group that uses the app, exercises (mindfulness, breathing), reminder systems, recording, reinforcement and monitoring will also be provided. It is estimated that a total of 112 participants (38 per group) will be necessary, and four evaluations will be carried out: T0 (pre-treatment), T1 (post-treatment, T2 (follow-up at three months) and T3 (follow-up at six months). months).

Hypothesis : The primary results that are expected to be obtained are a significant increase in the psychological flexibility of patients receiving treatment, with greater flexibility in the group receiving the combined intervention, evaluated with the AAQ-II. Furthermore, as secondary outcomes, it is expected to obtain significant improvements in anxiety and depression (HADS), quality of life (EORTC QLQ C-30), Fatigue (BFI), Insomnia (ISI) and post-traumatic growth (PTGI-SF).

Hypothesis: the efficacy of the ACT-based intervention in cancer patients may be increased if the benefits of using a modality that combines face-to-face and not face-to-face are added to it.

ELIGIBILITY:
The inclusion criteria for participants are:

* Men and women, aged between 18 and 70 years.
* Cancer diagnosis, stages I-III.
* Cancer type: Breast / Lung / Colorectal.
* Eligible for or currently receiving cancer treatment.
* Ability to be fluent in Spanish.
* Have a smartphone with daily access and basic smartphone / application management skills.
* Access to email account and internet.
* Not currently participating in another clinical trial.
* Not currently receiving other psychological treatment.

Exclusion criteria for participants in the trial:

* Men and women aged> 70 years.
* Diagnosis of cancer, stage IV or other types of cancer.
* Not eligible for treatment.
* Inability to handle himself fluently in Spanish.
* Not having a smartphone with daily access and basic smartphone / application skills.
* Not having access to an email account and the internet.
* Currently participating in another clinical trial.
* Currently receiving other psychological treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean of Psychological flexibility scores | Change of mean scores of psychological flexibility from baseline to immediately after intervention
  Acceptance and Action Questionnaire- II (AAQ-II). This instrument is designed to assess experiential avoidance and psychological inflexibility through 7 items that are answered with a Likert-type scale from 1 (never true) to 7 (always true) and a higher score indicates greater experiential avoidance (Bond et al., 2011).

SECONDARY OUTCOMES:
Mean of Anxiety and Depression scores | Change of mean scores of anxiety and depression from baseline to immediately after intervention
  Hospital Anxiety and Depression Scale (HADS). This scale is used to assess anxiety and depression in a hospital settings. It is made up of 14 items (7 for anxiety and 7 for depression), which are answered on a scale from 0 to 3, with maximum values of 21 in each of the subscales
Mean of Quality of Life scores using EORTC QLQ C-30 | Change of mean scores of the different subscales of quality of life from baseline to immediately after intervention
  EORTC QLQ C-30 (version 3), this is an instrument developed to assess the quality of life in cancer patients using 30 questions that refer to the quality of life experienced by the patient during the last week. The first twenty-eight items include questions about different symptoms and are answered on a scale that ranges from 1 (not at all) to 4 (a lot), while the last two ask patients about the perception of their global health and quality of life in a scale from 1 (terrible) to 7 (excellent). The different items are grouped into functional scales (physical / role / emotional / cognitive / social and global) and symptom scale (fatigue / nausea and vomiting / dyspnea / sleep problems / loss of appetite / constipation / diarrhea and financial impact ).
Mean of Fatigue scores | Change of mean scores of fatigue from baseline to immediately after intervention
  Brief Fatigue Inventory (BFI), is an instrument developed to assess fatigue in cancer patients that consists of 10 items with a Likert-type scale that assesses fatigue experienced in the last 24 hours from 0 (no fatigue) to 10 (worst fatigue imaginable). It also includes a scale to assess the degree to which fatigue has interfered with the patient's daily life in the last 24 hours, with a scale ranging from 0 (does not interfere) to 10 (completely inferred). The recommended cut-off points in cancer patients are: 1-3 (mild); 4-7 (moderate) and 8-10 (severe)
Mean of Insomnia scores | Change of mean scores of insomnia from baseline to immediately after intervention
  Insomnia Severity Index (ISI). This instrument is designed to assess the severity of insomnia experienced through 5 items that are scored on a scale from 0 (not at all) to 4 (very severe / very dissatisfied / very much). The sum of the scores given by the subject to the different items are added together and a total score is obtained that ranges from 0-28. The recommended cut-off points are as follows: 0-7 (absence of clinical insomnia), 8-14 (subclinical insomnia), 15-21 (moderate clinical insomnia), and 22-28 (severe clinical insomnia).
Mean in Post-Traumatic growth scores | Change of mean scores of post-traumatic growth from baseline to immediately after intervention
  Post-traumatic Growth Inventory-short version (PTGI-SF), is an instrument designed to evaluate the positive change that people who are subjected to a traumatic event may experience, using 10 items that respond to a Likert-type scale from 0 (no I have experienced that change) to 5 (I have experienced that change to a great extent), with higher scores showing greater positive change

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No
not applicable for this essay

REFERENCES:
- [Derived] Garcia-Torres F, Garcia-Carmona M, Gomez-Solis A, Jurado-Gonzalez F, Jablonski M, Jaen-Moreno MJ, Aranda E. Anxiety, depression, quality of life and the mediating role of psychological flexibility: A study on Spanish cancer patients. Sci Rep. 2025 Jul 2;15(1):22530. doi: 10.1038/s41598-025-06942-6. PMID 40595087
- [Derived] Garcia-Torres F, Gomez-Solis A, Rubio Garcia S, Castillo-Mayen R, Gonzalez Ruiz-Ruano V, Moreno E, Moriana JA, Luque-Salas B, Jaen-Moreno MJ, Cuadrado-Hidalgo F, Galvez-Lara M, Jablonski M, Rodriguez-Alonso B, Aranda E. Efficacy of a Combined Acceptance and Commitment Intervention to Improve Psychological Flexibility and Associated Symptoms in Cancer Patients: Study Protocol for a Randomized Controlled Trial. Front Psychol. 2022 May 18;13:871929. doi: 10.3389/fpsyg.2022.871929. eCollection 2022. PMID 35664159